CLINICAL TRIAL: NCT00842244
Title: A Phase 1 Study Of Axitinib In Combination With Cisplatin And Capecitabine In Patients With Advanced Gastric Cancer
Brief Title: Study Of Axitinib In Combination With Cisplatin And Capecitabine In Patients With Advanced Gastric Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4061055
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Results first posted 2012-03-26 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-10

CONDITIONS: Stomach Neoplasms; Advanced Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Axitinib; Capecitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: axitinib; Drug: capecitabine; Drug: cisplatin

INTERVENTIONS:
Drug: axitinib — Twice daily oral dose of axitinib continuously depending upon side effects observed. Starting dose is 5mg twice daily. Each 21 day cycle is repeated until progression of disease or unacceptable toxicity is observed.
Drug: capecitabine — Given orally twice daily for 14 days followed by 7 days of drug free period. Starting dose is 1000mg/m^2 twice daily. Each 21 day cycle is repeated until progression of disease or unacceptable toxicity is observed.
Drug: cisplatin — Given through a vein on Day 1 of every 21 days. Each 21 day cycle is repeated until progression of disease or unacceptable toxicity is observed. The starting dose is 80 mg/m^2 on day 1.

SUMMARY:
The purpose of this study is to determine the safe and tolerable dose of axitinib given together with cisplatin and capecitabine in patients with advanced gastric cancer who have not received prior chemotherapy for their advanced cancer.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of stomach cancer
* advanced stomach cancer of stage IV
* adequate blood chemistry, blood counts and kidney function
* willing to participate to study requirements and sign an informed consent document

Exclusion Criteria:

* prior chemotherapy for stomach cancer in its advanced stage
* excessive toxicities related to prior therapies
* pregnant or breastfeeding patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-04; Primary Completion 2009-12 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- Japan (2):
  - Pfizer Investigational Site, Kashiwa, Chiba
  - Pfizer Investigational Site, Yufu, Oita Prefecture
- South Korea (3):
  - Pfizer Investigational Site, Goyang-si, Gyeonggi-do
  - Pfizer Investigational Site, Seongnam-si, Gyeonggi-do
  - Pfizer Investigational Site, Seoul

REFERENCES:
- [Derived] Oh DY, Doi T, Shirao K, Lee KW, Park SR, Chen Y, Yang L, Valota O, Bang YJ. Phase I Study of Axitinib in Combination with Cisplatin and Capecitabine in Patients with Previously Untreated Advanced Gastric Cancer. Cancer Res Treat. 2015 Oct;47(4):687-96. doi: 10.4143/crt.2014.225. Epub 2015 Feb 12. PMID 25687867
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4061055&StudyName=Study%20Of%20Axitinib%20In%20Combination%20With%20Cisplatin%20And%20Capecitabine%20In%20Patients%20With%20Advanced%20Gastric%20Cancer

RESULTS

PARTICIPANT FLOW:
Groups:
- Axitinib + Capecitabine + Cisplatin: Axitinib (AG-013736) 5 milligram (mg) tablet orally twice daily in cycles of 21 days, capecitabine 1000 mg per square meter (mg/m^2) tablet orally twice daily from Day 1 to 14 of each cycle and cisplatin 80 mg/m^2 infusion over 2 hours (hrs) on Day 1 of each cycle, in cycles of 21 days. Participants enrolled in pharmacokinetic (PK) expansion cohort at maximum tolerated dose (MTD) received axitinib (AG-013736) 5 mg orally twice daily starting from Day -3 to Day 18 in Cycle 1 (21 days cycle) and thereafter axitinib (AG-013736) 5 mg orally twice daily starting from Cycle 2 Day 2, capecitabine 1000 mg/m^2 tablet orally twice daily from Day 1 to 14 and cisplatin 80 mg/m^2 infusion over 2 hrs on Day 1 of each cycle, in cycles of 21 days.
Period: Overall Study
Arm/Group | Axitinib + Capecitabine + Cisplatin
Started | 22
Completed | 1
Not Completed | 21
Not completed — Death | 3
Not completed — Withdrawal by Subject | 1
Not completed — Other | 17

BASELINE CHARACTERISTICS:
Arm/Group | Axitinib + Capecitabine + Cisplatin
Number analyzed (Participants) | 22
Age Continuous [Mean (Standard Deviation); unit: years] | 59.3 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Cycle 1 Dose-limiting Toxicities (DLTs)
Description: DLT = Grade (GR) 2 proteinuria; GR3 nonhematological toxicity (NHT) (excluding alopecia and those that can be controlled with appropriate treatment) for greater than or equal to (>=)7 days, GR3 thrombocytopenia with active bleeding; GR >=3 febrile neutropenia (NP) or NP infection; GR 3 or 4 nausea, vomiting or diarrhea despite anti-emetics, anti-diarrheals; GR4 NHT, thrombocytopenia, NP for >=7 days; >= 1/2 teaspoon per day hemoptysis; any treatment related toxicity with >3 consecutive days of capecitabine or 5 consecutive days of axitinib missed doses per cycle; delayed toxicity recovery >14 days.
Time Frame: Baseline up to Day 21 of Cycle 1
Population: DLT analysis set: participants who received first cycle of study treatment and did not temporarily or permanently discontinue or miss more than 5 consecutive days of axitinib (AG-13736) or more than 3 consecutive days of capecitabine for reasons other than DLTs within first cycle.
Measure: Number; unit: participants
Groups:
- Axitinib + Capecitabine + Cisplatin (MTD Determination): Axitinib (AG-013736) 5 mg tablet orally twice daily in cycles of 21 days, capecitabine 1000 mg/m^2 tablet orally twice daily from Day 1 to 14 of each cycle and cisplatin 80 mg/m^2 infusion over 2 hrs on Day 1 of each cycle, in cycles of 21 days.
Arm/Group | Axitinib + Capecitabine + Cisplatin (MTD Determination)
Number analyzed (Participants) | 12
participants | 3

2. Other Pre Specified Outcome: Maximum Tolerated Dose (MTD) of Axitinib (AG-013736) in Combination With Cisplatin and Capecitabine
Description: MTD = highest dose at which no more than 30 percent (%) of 12 participants experience DLT during Cycle 1. DLT = GR2 proteinuria; GR3 NHT (excluding alopecia and those that can be controlled with appropriate treatment)for >=7 days, GR3 thrombocytopenia with active bleeding; GR >=3 febrile NP/NP infection; GR 3 or 4 nausea, vomiting or diarrhea despite anti-emetics, anti-diarrheals; GR4 NHT, thrombocytopenia, NP for >=7 days; >= 1/2 teaspoon per day hemoptysis; any treatment-related toxicity with >3 consecutive days of capecitabine or 5 consecutive days of axitinib missed doses per cycle; delayed toxicity recovery >14 days.
Time Frame: Baseline up to Day 21 of Cycle 1
Population: as for outcome 1
Measure: Number; unit: mg
Arm/Group | Axitinib + Capecitabine + Cisplatin (MTD Determination)
Number analyzed (Participants) | 12
mg | 5

3. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Axitinib, Capecitabine, Capecitabine's Metabolites and Cisplatin
Description: Cmax for axitinib in absence of chemotherapy (axitinib alone) was evaluated on Cycle 1 Day -1 and in combination with chemotherapy on Cycle 1 Day 1. Cmax for cisplatin (assessed by estimating total platinum in plasma ultrafiltrate), capecitabine and capecitabine's metabolites (5-fluorouracil [5-FU], 5-deoxy-5-fluorouridine [5-DFUR] and 5-deoxy-5-fluorocytidine [5-DFC]) in presence of steady-state axitinib were evaluated on Cycle 1 Day 1 and in absence of axitinib (cisplatin/capecitabine alone) on Cycle 2 Day 1. Results for axitinib were normalized to axitinib 5 mg dose, results for capecitabine and its metabolites (5-FU, 5-DFUR and 5-DFC) were normalized to Cycle 1 Day 1 capecitabine dose and results for cisplatin were normalized to Cycle 1 Day 1 cisplatin dose.
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 6, 8 hrs post-axitinib dose on Cycle 1 (C1) Day -1 (D-1), C1D1; 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 4, 6, 8 hrs post-capecitabine dose C1D1, C2D1; 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8 hrs post-cisplatin infusion start C1D1, C2D1
Population: Pharmacokinetic parameter analysis set included all treated participants who had at least 1 estimated pharmacokinetic parameter of primary interest. Here, 'n' signifies those participants who were evaluable for specified study drug's PK parameter alone or in combination.
Measure: Geometric Mean (95% Confidence Interval); unit: nanogram/milliliter (ng/mL)
Groups:
- Axitinib + Capecitabine + Cisplatin (PK Expansion Cohort): Participants enrolled in PK expansion cohort at MTD received axitinib (AG-013736) 5 mg orally twice daily starting from Day -3 to Day 18 in Cycle 1 (21 days cycle) and thereafter axitinib (AG-013736) 5 mg orally twice daily starting from Cycle 2 Day 2, capecitabine 1000 mg/m^2 tablet orally twice daily from Day 1 to 14 and cisplatin 80 mg/m^2 infusion over 2 hrs on Day 1 of each cycle, in cycles of 21 days.
Arm/Group | Axitinib + Capecitabine + Cisplatin (PK Expansion Cohort)
Number analyzed (Participants) | 10
nanogram/milliliter (ng/mL)
  Axitinib alone (n = 10) | 16.11 [9.94 to 26.10]
  Axitinib in combination with chemotherapy (n = 10) | 24.33 [15.01 to 39.43]
  Capecitabine alone (n = 8) | 5255.62 [3155.36 to 8753.85]
  Capecitabine in presence of axitinib (n = 8) | 2274.80 [1365.74 to 3788.95]
  5-FU alone (n = 8) | 220.49 [132.31 to 367.44]
  5-FU in presence of axitinib (n = 8) | 90.97 [54.59 to 151.59]
  5-DFUR alone (n = 8) | 5791.81 [3871.80 to 8663.95]
  5-DFUR in presence of axitinib (n = 8) | 3017.27 [2017.03 to 4513.52]
  5-DFC alone (n = 8) | 5891.29 [4416.64 to 7858.31]
  5-DFC in presence of axitinib (n = 8) | 3227.57 [2419.68 to 4305.21]
  Cisplatin alone (n = 8) | 1665.27 [1407.48 to 1970.26]
  Cisplatin in presence of axitinib (n = 8) | 1865.07 [1576.36 to 2206.66]

4. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) for Axitinib, Capecitabine, Capecitabine's Metabolites and Cisplatin
Description: Tmax for axitinib in absence of chemotherapy (axitinib alone) was evaluated on Cycle 1 Day -1 and in combination with chemotherapy on Cycle 1 Day 1. Tmax for cisplatin (assessed by estimating total platinum in plasma ultrafiltrate), capecitabine and capecitabine's metabolites (5-FU, 5-DFUR and 5-DFC) in presence of steady-state axitinib were evaluated on Cycle 1 Day 1 and in absence of axitinib (cisplatin/capecitabine alone) on Cycle 2 Day 1.
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 6, 8 hrs post-axitinib dose on C1D-1, C1D1; 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 4, 6, 8 hrs post-capecitabine dose C1D1, C2D1; 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8 hrs post-cisplatin infusion start C1D1, C2D1
Population: as for outcome 3
Measure: Median (Full Range); unit: hrs
Arm/Group | Axitinib + Capecitabine + Cisplatin (PK Expansion Cohort)
Number analyzed (Participants) | 10
hrs
  Axitinib alone (n = 10) | 3.98 [0.00 to 7.97]
  Axitinib in combination with chemotherapy (n = 10) | 4.00 [1.00 to 6.00]
  Capecitabine alone (n = 8) | 2.45 [0.50 to 4.00]
  Capecitabine in presence of axitinib (n = 8) | 3.12 [0.50 to 4.02]
  5-FU alone (n = 8) | 2.50 [0.50 to 4.07]
  5-FU in presence of axitinib (n = 8) | 2.62 [0.50 to 4.02]
  5-DFUR alone (n = 8) | 2.50 [0.50 to 4.07]
  5-DFUR in presence of axitinib (n = 8) | 2.62 [0.97 to 4.02]
  5-DFC alone (n = 8) | 2.50 [0.50 to 4.07]
  5-DFC in presence of axitinib (n = 8) | 3.09 [0.50 to 4.02]
  Cisplatin alone (n = 8) | 2.00 [1.00 to 2.20]
  Cisplatin in presence of axitinib (n = 8) | 1.02 [0.97 to 2.33]

5. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for Capecitabine, Capecitabine's Metabolites and Cisplatin
Description: Area under the plasma concentration time-curve from zero to the last measurable concentration (AUClast). AUClast for cisplatin (assessed by estimating total platinum in plasma ultrafiltrate), capecitabine and capecitabine's metabolites (5-FU, 5-DFUR, 5-DFC) in presence of steady-state axitinib were evaluated on Cycle 1 Day 1 and in absence of axitinib (cisplatin/capecitabine alone) on Cycle 2 Day 1. Results for capecitabine and its metabolites (5-FU, 5-DFUR and 5-DFC) were normalized to Cycle 1 Day 1 capecitabine dose and results for cisplatin were normalized to Cycle 1 Day 1 cisplatin dose.
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 4, 6, 8 hrs post-capecitabine dose C1D1, C2D1; 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8 hrs post-cisplatin infusion start C1D1, C2D1
Population: Pharmacokinetic parameter analysis set included all treated participants who had at least 1 estimated pharmacokinetic parameter of primary interest. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Geometric Mean (95% Confidence Interval); unit: nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | Axitinib + Capecitabine + Cisplatin (PK Expansion Cohort)
Number analyzed (Participants) | 8
nanogram*hour/milliliter (ng*hr/mL)
  Capecitabine alone | 7109.59 [4525.07 to 11170.27]
  Capecitabine in presence of axitinib | 4194.97 [2669.99 to 6590.95]
  5-FU alone | 332.37 [238.03 to 464.12]
  5-FU in presence of axitinib | 176.81 [126.62 to 246.89]
  5-DFUR alone | 9996.55 [8183.62 to 12211.10]
  5-DFUR in presence of axitinib | 6683.33 [5471.27 to 8163.90]
  5-DFC alone | 10820.14 [8838.29 to 13246.37]
  5-DFC in presence of axitinib | 7983.14 [6520.93 to 9773.23]
  Cisplatin alone | 3814.93 [3463.52 to 4202.00]
  Cisplatin in presence of axitinib | 3951.57 [3587.57 to 4352.50]

6. Secondary Outcome: Area Under the Curve From Time Zero to 24 Hours [AUC (0-24)] for Axitinib
Description: AUC (0-24) = Area under the plasma concentration versus time curve from time zero (pre-dose) to 24 hours. AUC (0-24) for axitinib in absence of chemotherapy (axitinib alone) was evaluated on Cycle 1 Day -1 and in combination with chemotherapy on Cycle 1 Day 1. Results for axitinib were normalized to axitinib 5 mg dose.
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 6, 8 hrs post-axitinib dose on C1D-1, C1D1
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: ng*hr/mL
Arm/Group | Axitinib + Capecitabine + Cisplatin (PK Expansion Cohort)
Number analyzed (Participants) | 9
ng*hr/mL
  Axitinib alone | 206.20 [109.20 to 389.36]
  Axitinib in combination with chemotherapy | 265.89 [140.81 to 502.08]

7. Secondary Outcome: Area Under the Curve From Time Zero Extrapolated to Infinite Time [AUC (0 - ∞)] for Axitinib, Capecitabine, Capecitabine's Metabolites and Cisplatin
Description: AUC (0 - ∞) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) extrapolated to infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞). AUC (0 - ∞) for axitinib in absence of chemotherapy (axitinib alone) was evaluated on Cycle 1 Day -1 and in combination with chemotherapy on Cycle 1 Day 1. AUC (0 - ∞) for cisplatin (assessed by estimating total platinum in plasma ultrafiltrate), capecitabine and capecitabine's metabolites (5-FU, 5-DFUR and 5-DFC) in presence of steady-state axitinib were evaluated on Cycle 1 Day 1 and in absence of axitinib (cisplatin/capecitabine alone) on Cycle 2 Day 1. Results for axitinib were normalized to axitinib 5 mg dose, results for capecitabine and its metabolites (5-FU, 5-DFUR and 5-DFC) were normalized to Cycle 1 Day 1 capecitabine dose and results for cisplatin were normalized to Cycle 1 Day 1 cisplatin dose.
Time Frame: as for outcome 4
Population: Pharmacokinetic parameter analysis set. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. Here, 'n' signifies those participants who were evaluable for specified study drug's PK parameter alone or in combination.
Measure: Geometric Mean (95% Confidence Interval); unit: ng*hr/mL
Arm/Group | Axitinib + Capecitabine + Cisplatin (PK Expansion Cohort)
Number analyzed (Participants) | 9
ng*hr/mL
  Axitinib alone (n = 9) | 147.04 [70.79 to 305.42]
  Axitinib in combination with chemotherapy (n = 9) | 156.00 [75.10 to 324.02]
  Capecitabine alone (n = 6) | 7140.62 [4197.86 to 12146.29]
  Capecitabine in presence of axitinib (n = 6) | 4213.72 [2477.18 to 7167.60]
  5-FU alone (n = 3) | 337.85 [198.44 to 575.20]
  5-FU in presence of axitinib (n = 3) | 261.95 [153.86 to 445.98]
  5-DFUR alone (n = 4) | 9568.70 [6772.04 to 13520.28]
  5-DFUR in presence of axitinib (n = 4) | 6966.07 [4930.09 to 9842.84]
  5-DFC alone (n = 5) | 11587.97 [7974.00 to 16839.87]
  5-DFC in presence of axitinib (n = 5) | 7787.39 [5358.71 to 11316.78]
  Cisplatin alone (n = 7) | 3979.07 [3577.60 to 4425.59]
  Cisplatin in presence of axitinib (n = 7) | 3990.34 [3587.74 to 4438.12]

8. Secondary Outcome: Plasma Decay Half-Life (t1/2) for Axitinib, Capecitabine, Capecitabine's Metabolites and Cisplatin
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half. Plasma decay half life for axitinib in absence of chemotherapy (axitinib alone) was evaluated on Cycle 1 Day -1 and in combination with chemotherapy on Cycle 1 Day 1. Plasma decay half life for cisplatin (assessed by estimating total platinum in plasma ultrafiltrate), capecitabine and capecitabine's metabolites (5-FU, 5-DFUR and 5-DFC) in presence of steady-state axitinib were evaluated on Cycle 1 Day 1 and in absence of axitinib (cisplatin/capecitabine alone) on Cycle 2 Day 1.
Time Frame: as for outcome 4
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hrs
Arm/Group | Axitinib + Capecitabine + Cisplatin (PK Expansion Cohort)
Number analyzed (Participants) | 9
hrs
  Axitinib alone (n = 9) | 5.76 (3.665)
  Axitinib in combination with chemotherapy (n = 9) | 3.50 (1.869)
  Capecitabine alone (n = 6) | 0.71 (0.441)
  Capecitabine in presence of axitinib (n = 6) | 0.89 (0.520)
  5-FU alone (n = 3) | 1.11 (0.455)
  5-FU in presence of axitinib (n = 3) | 1.05 (0.506)
  5-DFUR alone (n = 4) | 0.96 (0.400)
  5-DFUR in presence of axitinib (n = 4) | 0.77 (0.125)
  5-DFC alone (n = 5) | 0.98 (0.499)
  5-DFC in presence of axitinib (n = 5) | 0.78 (0.147)
  Cisplatin alone (n = 7) | 1.25 (0.095)
  Cisplatin in presence of axitinib (n = 7) | 1.61 (0.772)

9. Secondary Outcome: Apparent Oral Clearance (CL/F) for Axitinib, Capecitabine and Capecitabine's Metabolites
Description: Clearance (CL) of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed (F). Clearance is defined as the volume of blood from which drug can be completely removed per unit of time. CL/F for axitinib in absence of chemotherapy (axitinib alone) was evaluated on Cycle 1 Day -1 and in combination with chemotherapy on Cycle 1 Day 1. CL/F for capecitabine in presence of steady-state axitinib was evaluated on Cycle 1 Day 1 and in absence of axitinib (capecitabine alone) on Cycle 2 Day 1.
Time Frame: 0 (pre-dose), 1, 2, 3, 4, 6, 8 hrs post-axitinib dose on C1D-1, C1D1; 0 (pre-dose), 0.25, 0.5, 1, 2, 3, 4, 6, 8 hrs post-capecitabine dose on C1D1, C2D1
Population: Pharmacokinetic parameter analysis set. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. 'n' = participants evaluable for specified study drug's PK parameter alone or in combination. Results are not reported for capecitabine metabolites because CL/F could not be accurately estimated.
Measure: Geometric Mean (95% Confidence Interval); unit: Liter/hr
Arm/Group | Axitinib + Capecitabine + Cisplatin (PK Expansion Cohort)
Number analyzed (Participants) | 9
Liter/hr
  Axitinib alone (n = 9) | 48.55 [25.71 to 91.70]
  Axitinib in combination with chemotherapy (n = 9) | 37.69 [19.96 to 71.19]
  Capecitabine alone (n = 6) | 217.60 [118.45 to 399.74]
  Capecitabine in presence of axitinib (n = 6) | 368.47 [200.58 to 676.89]

10. Secondary Outcome: Clearance (CL) for Cisplatin
Description: Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood. It is defined as the volume of blood from which drug can be completely removed per unit of time. Clearance for cisplatin (assessed by estimating total platinum in plasma ultrafiltrate) in presence of steady-state axitinib was evaluated on Cycle 1 Day 1 and in absence of axitinib (cisplatin alone) on Cycle 2 Day 1.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8 hrs post-cisplatin infusion start on C1D1, C2D1
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Liter/hr
Arm/Group | Axitinib + Capecitabine + Cisplatin (PK Expansion Cohort)
Number analyzed (Participants) | 7
Liter/hr
  Cisplatin alone | 30.94 [26.03 to 36.77]
  Cisplatin in presence of axitinib | 32.50 [27.35 to 38.63]

11. Secondary Outcome: Apparent Volume of Distribution (Vz/F) for Axitinib, Capecitabine and Capecitabine's Metabolites
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Vz/F is influenced by the fraction absorbed. Vz/F for axitinib in absence of chemotherapy (axitinib alone) was evaluated on Cycle 1 Day -1 and in combination with chemotherapy on Cycle 1 Day 1. Vz/F for capecitabine in presence of steady-state axitinib was evaluated on Cycle 1 Day 1 and in absence of axitinib (capecitabine alone) on Cycle 2 Day 1.
Time Frame: as for outcome 9
Population: Pharmacokinetic parameter analysis set. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. 'n' = participants evaluable for specified study drug's PK parameter alone or in combination. Results are not reported for capecitabine metabolites because Vz/F could not be accurately estimated.
Measure: Geometric Mean (95% Confidence Interval); unit: Liter
Arm/Group | Axitinib + Capecitabine + Cisplatin (PK Expansion Cohort)
Number analyzed (Participants) | 9
Liter
  Axitinib alone (n = 9) | 344.87 [202.24 to 588.09]
  Axitinib in combination with chemotherapy (n = 9) | 171.83 [100.77 to 293.01]
  Capecitabine alone (n = 6) | 190.94 [89.08 to 409.30]
  Capecitabine in presence of axitinib (n = 6) | 425.00 [198.27 to 911.02]

12. Secondary Outcome: Volume of Distribution (Vz) for Cisplatin
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Clearance for cisplatin (assessed by estimating total platinum in plasma ultrafiltrate) in presence of steady-state axitinib was evaluated on Cycle 1 Day 1 and in absence of axitinib (cisplatin alone) on Cycle 2 Day 1.
Time Frame: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8 hrs post-cisplatin infusion start on C1D1, C2D1
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Liter
Arm/Group | Axitinib + Capecitabine + Cisplatin (PK Expansion Cohort)
Number analyzed (Participants) | 7
Liter
  Cisplatin alone | 55.35 [41.12 to 74.51]
  Cisplatin in presence of axitinib | 70.32 [52.24 to 94.66]

13. Secondary Outcome: Drug Metabolizing Enzyme Genotyping
Description: Genetic variants of uridine diphosphate (UDP)- glucuronosyl transferase 1A1 (UGT1A1) gene which were assessed for genotyping included UGT1A1*60, UGT1A1-3156, UGT1A1 Promoter thymine adenine (TA) repeat (UGT1A1*28, UGT1A1*36, UGT1A1*37), UGT1A1*6 and UGT1A1*27.
Time Frame: Day 1 of Cycle 1
Population: Results are not reported because data was reported in individual participant listing but not statistically summarized for the analysis.
Groups:
- Axitinib + Capecitabine + Cisplatin: Axitinib (AG-013736) 5 milligram (mg) tablet orally twice daily in cycles of 21 days, capecitabine 1000 mg per square meter (mg/m^2) tablet orally twice daily from Day 1 to 14 of each cycle and cisplatin 80 mg/m^2 infusion over 2 hours (hrs) on Day 1 of each cycle, in cycles of 21 days. Participants enrolled in Pharmacokinetic (PK) expansion cohort at MTD received axitinib (AG-013736) 5 mg orally twice daily starting from Day -3 to Day 18 in Cycle 1 (21 days cycle) and thereafter axitinib (AG-013736) 5 mg orally twice daily starting from Cycle 2 Day 2, capecitabine 1000 mg/m^2 tablet orally twice daily from Day 1 to 14 and cisplatin 80 mg/m^2 infusion over 2 hrs on Day 1 of each cycle, in cycles of 21 days.
Arm/Group | Axitinib + Capecitabine + Cisplatin
Number analyzed (Participants) | 0

14. Secondary Outcome: Percentage of Participants With Objective Response (OR)
Description: Number of participants with objective response based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed response are those that persist on repeat imaging study at least 4 weeks after initial documentation of response. CR are those with disappearance of all target lesions. PR are those with at least 30 percent (%) decrease in sum of the longest dimensions of target lesions taking the baseline sum of the longest dimensions as a reference.
Time Frame: Baseline up to disease progression or withdrawal, assessed on Day 21 of every other cycle starting from Cycle 2 up to Day 784
Population: Efficacy analysis set included all enrolled participants who received at least 1 dose of study medication, had measurable disease at baseline (according to RECIST criteria version 1.0), and had at least 1 tumor assessment during study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Axitinib + Capecitabine + Cisplatin
Number analyzed (Participants) | 22
percentage of participants | 36.36 [17.2 to 59.34]

15. Secondary Outcome: Duration of Response (DR)
Description: Time in months from the first documentation of objective tumor response to objective tumor progression or death due to any cause. Duration of tumor response was calculated as (the date of the first documentation of objective tumor progression or death minus the date of the first CR or PR that was subsequently confirmed plus 1) divided by 30.4. DR was calculated for the subgroup of participants with a confirmed objective tumor response. CR = disappearance of all target lesions. PR = at least 30% decrease in sum of the longest dimensions of target lesions taking the baseline sum of the longest dimensions as a reference.
Time Frame: as for outcome 14
Population: Analysis set included a subset of efficacy analysis set who had confirmed objective tumor response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axitinib + Capecitabine + Cisplatin
Number analyzed (Participants) | 8
months | 9.07 [6.44 to 20.20]

16. Secondary Outcome: Progression-Free Survival (PFS)
Description: Time in months from start of study treatment to first documentation of objective tumor progression or death due to any cause. PFS was calculated as (first event date minus the date of first dose of study medication plus 1) divided by 30.4. Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD]), or from adverse event (AE) data (where the outcome was "Death"). PD was a>=20% increase in sum of the longest dimensions of target lesions taking as a reference the smallest sum of the longest dimensions recorded since the treatment started, or the appearance of 1 or more new lesions.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axitinib + Capecitabine + Cisplatin
Number analyzed (Participants) | 22
months | 3.75 [2.92 to 9.40]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Axitinib + Capecitabine + Cisplatin
Serious Adverse Events (participants affected / at risk) | 12/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib + Capecitabine + Cisplatin (N=22)
Bradycardia (Cardiac disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 1
Headache (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Aortic aneurysm rupture (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Acute prerenal failure (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib + Capecitabine + Cisplatin (N=22)
Anaemia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 14
Thrombocytopenia (Blood and lymphatic system disorders) | 12
Tinnitus (Ear and labyrinth disorders) | 2
Hypothyroidism (Endocrine disorders) | 10
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 6
Cheilitis (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 9
Diarrhoea (Gastrointestinal disorders) | 12
Dyspepsia (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 17
Periodontitis (Infections and infestations) | 2
Stomatitis (Gastrointestinal disorders) | 16
Vomiting (Gastrointestinal disorders) | 7
Asthenia (General disorders) | 4
Fatigue (General disorders) | 17
Mucosal inflammation (General disorders) | 2
Oedema (General disorders) | 2
Pyrexia (General disorders) | 2
Oral candidiasis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 3
Alanine aminotransferase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 2
Blood creatinine increased (Investigations) | 3
Haemoglobin decreased (Investigations) | 3
Neutrophil count decreased (Investigations) | 2
Weight decreased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 20
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Dysgeusia (Nervous system disorders) | 3
Headache (Nervous system disorders) | 4
Neuropathy peripheral (Nervous system disorders) | 4
Insomnia (Psychiatric disorders) | 2
Proteinuria (Renal and urinary disorders) | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 12
Hiccups (Respiratory, thoracic and mediastinal disorders) | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 2
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 12
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 3
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 16
Hypotension (Vascular disorders) | 3
Abdominal discomfort (Gastrointestinal disorders) | 2

LIMITATIONS AND CAVEATS:
AUC (0-24) was evaluated and reported for axitinib instead of AUClast as AUC0-24 was a more appropriate measure of steady-state exposure for this drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.